CLINICAL TRIAL: NCT05329935
Title: Congenital Athymia Patient Registry of RETHYMIC
Brief Title: Congenital Athymia Patient Registry
Status: Recruiting | Type: Observational
Sponsor: Sumitomo Pharma Switzerland GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: RVT-802-4001
Record Dates: First submitted 2022-03-24; First posted 2022-04-15 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Complete DiGeorge Anomaly; Complete DiGeorge Syndrome; Congenital Athymia
Keywords: Congenital Athymia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Main cohort: All eligible patients
  Interventions: Biological: Cultured Thymus Tissue
- Secondary cohort: All eligible patients who survived 1 year post treatment
  Interventions: Biological: Cultured Thymus Tissue

INTERVENTIONS:
Biological: Cultured Thymus Tissue — Product will be surgically administered into the quadriceps
  Other Names: RETHYMIC; allogeneic cultured thymus tissue-agdc

SUMMARY:
This Congenital Athymia Patient Registry is an observational exposure-based registry study. It uses a prospective cohort design to follow patients who have been treated with RETHYMIC.

Clinical studies conducted with investigational RETHYMIC showed that treatment can result in immune reconstitution and prolong life. This treatment-based registry is being conducted to learn more about the reconstitution process following treatment and the impact of treatment on longer-term survival and the occurrence of adverse events of special interest (AESI).

DETAILED DESCRIPTION:
This Congenital Athymia Patient Registry is an observational exposure-based registry study. It uses a prospective cohort design to follow patients who have been treated with RETHYMIC.

Clinical studies conducted with investigational RETHYMIC showed that treatment can result in immune reconstitution and prolong life. This treatment-based registry is being conducted to learn more about the reconstitution process following treatment and the impact of treatment on longer-term survival and the occurrence of adverse events of special interest (AESI).

Currently, there is a single site where patients are being treated with RETHYMIC. The Investigator will be responsible for recruiting patients who have recently had (i.e., within the past 60 days) or are scheduled to have this treatment within 30 days and obtaining signed informed consent (and assent as applicable). The Investigator will collect baseline medical history and clinical data information for each enrolled subject. The start of follow-up (day 1) begins on the day following treatment surgery. Clinical data and flow cytometry test results (when conducted) will be abstracted from the medical records by Clinical Staff at baseline and during follow-up at predefined intervals.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients diagnosed with Congenital Athymia:

  * Who are scheduled for implantation with RETHYMIC within the next 30 days, or who were treated with RETHYMIC within the previous 60 days.
  * Who have provided written informed consent directly, or written informed consent has been provided by the patient, the parent, or legal guardian.

Exclusion Criteria:

* Written informed consent cannot be obtained.

Ages: 0 Years to 21 Years | Sex: All
Age Groups: Child, Adult
Study Population: Pediatric patients diagnosed with Congenital Athymia:
  • Who are scheduled for implantation with RETHYMIC within the next 30 days, or who were treated with RETHYMIC within the previous 60 days.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Vital Status | 12 months post treatment with RETHYMIC.
Flow cytometry including total and naïve CD3, CD4, and CD8 counts | Immediately after the intervention/procedure/surgery

SECONDARY OUTCOMES:
AESI classified by MedDRA coding, severity and grade | Immediately after the intervention/procedure/surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University School of Medicine, Durham, North Carolina, United States

REFERENCES:
- [Background] RETHYMIC US Prescribing Information, 2021.